CLINICAL TRIAL: NCT06285240
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Assess the Safety, Tolerability, and Pharmacokinetics of MK-1167 Administered to Patients With Alzheimer's Disease Receiving Stable Donepezil Treatment
Brief Title: Efficacy and Safety of MK-1167 in Participants With Alzheimer's Disease Dementia Taking Stable Donepezil Treatment (MK-1167-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1167-007; MK-1167-007 (Other: MSD)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: Panel A participants will receive a loading dose of MK-1167 6mg or matching Placebo on Days 1 to 7 followed by once daily (QD) dosing of MK-1167 3mg or matching Placebo for 14 consecutive days (Days 8 to 21). Panel B participants will receive QD dosing of MK-1167 6mg or matching Placebo for Days 1 to 31. Panel B will be initiated following review of safety and tolerability data from Panel A.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Panel A: MK-1167 + Donepezil 10mg QD (Experimental): Participants receive 6mg MK-1167 oral loading doses once daily (QD) Days 1 to 7, followed by 3mg MK-1167 oral maintenance doses QD Days 8 to 21. Participants also receive 10mg oral Donepezil on Days -3 to 21.
  Interventions: Drug: MK-1167; Drug: Donepezil
- Panel A: Placebo to MK-1167 + Donepezil 10mg QD (Placebo Comparator): Participants receive dose matched placebo to MK-1167 oral QD from Days 1 to 21. Participants also receive 10mg oral Donepezil QD on Days -3 to 21.
  Interventions: Drug: Donepezil; Drug: Placebo
- Panel B: MK-1167 6mg QD + Donepezil 10mg QD (Experimental): Participants receive 6mg MK-1167 oral doses QD Days 1 to 31. Participants also receive 10mg oral Donepezil on Days -3 to 31.
  Interventions: Drug: MK-1167; Drug: Donepezil
- Panel B: Placebo to MK-1167 + Donepezil 10mg QD (Placebo Comparator): Participants receive dose matched placebo to MK-1167 oral QD from Days 1 to 31. Participants also receive 10mg oral Donepezil QD on Days -3 to 31.
  Interventions: Drug: Donepezil; Drug: Placebo

INTERVENTIONS:
Drug: MK-1167 — 1 mg and 5 mg oral capsules
  Arms: Panel A: MK-1167 + Donepezil 10mg QD; Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Drug: Donepezil — 10 mg oral tablets
Drug: Placebo — MK-1167 matching placebo administered oral capsules
  Arms: Panel A: Placebo to MK-1167 + Donepezil 10mg QD; Panel B: Placebo to MK-1167 + Donepezil 10mg QD

SUMMARY:
The main purpose of this study is to assess the safety and efficacy of MK-1167 administered to participants with Alzheimer's Disease (AD) receiving stable Donepezil treatment.

ELIGIBILITY:
Inclusion Criteria:

* Reports a history of cognitive and functional decline with gradual onset and slow progression for at least 1 year before Screening, that is either corroborated by an informant who knows the subject well or is documented in medical records
* Meets the criteria for a diagnosis of probable Alzheimer's disease (AD) based on the National Institute of Neurological and Communicative Disorders - Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable AD
* Is receiving donepezil 10 mg daily for symptomatic treatment of cognitive impairment associated with AD. The dose level must be stable for at least 2 months prior to Screening. If receiving donepezil via a transdermal system (ie, patch), it should be a 10-mg/day dose and should switch prescription to a 10-mg oral daily dose, before enrollment
* Has a reliable and competent trial partner/caregiver who has a close relationship with the participant, has face-to-face contact at least 3 days a week for a minimum of 6 waking hours a week, and is willing to accompany the participant, if desired, to study visits

Exclusion Criteria:

* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases that are not under medical control over the past 2 months.
* Has evidence of a clinically relevant or unstable psychiatric disorder, based on DSM-5 criteria, or has a history of clinically significant psychiatric disorder in the last 5 years. Generalized anxiety disorder, and/or insomnia under good control for ≥ 2 months on stable medical therapy may not be exclusionary.
* History of cancer (malignancy). Participants with adequately treated disease deemed as "cured," or who, in the opinion of the study investigator, are highly unlikely to sustain a recurrence for the duration of the study, may be enrolled at the discretion of the investigator and Sponsor.
* History of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or nonprescription drugs or food.
* Had a major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study intervention, throughout the study, until the poststudy visit. There may be certain protocol-specified medications that are permitted.
* The participant is a smoker and/or has used nicotine or nicotine-containing products (eg, nicotine patch and electronic cigarette) within 3 months of screening.
* Consumes greater than 3 servings of alcoholic beverages per day. Participants who consume 4 servings of alcoholic beverages per day may be enrolled at the discretion of the investigator.
* The participant is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Velocity Clinical Research, Hallandale Beach ( Site 0001), Hallandale, Florida
  - CenExel iResearch, LLC ( Site 0003), Decatur, Georgia
  - CenExel iResearch, LLC ( Site 0004), Savannah, Georgia

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants
Groups:
- Panel A: MK-1167 + Donepezil 10mg QD: Participants received 6mg MK-1167 oral loading doses once daily (QD) Days 1 to 7, followed by 3mg MK-1167 oral maintenance doses QD Days 8 to 21. Participants also received 10mg oral Donepezil on Days -3 to 21.
- Panel A: Placebo to MK-1167 + Donepezil 10mg QD: Participants received dose matched placebo to MK-1167 oral QD from Days 1 to 21. Participants also received 10mg oral Donepezil QD on Days-3 to 21.
- Panel B: MK-1167 6mg QD + Donepezil 10mg QD: Participants received 6mg MK-1167 oral doses QD Days 1 to 31. Participants also received 10mg oral Donepezil on Days -3 to 31.
- Panel B: Placebo to MK-1167 + Donepezil 10mg QD: Participants received dose matched placebo to MK-1167 oral QD from Days 1 to 31. Participants also received 10mg oral Donepezil QD on Days-3 to 31.
Period: Overall Study
Arm/Group | Panel A: MK-1167 + Donepezil 10mg QD | Panel A: Placebo to MK-1167 + Donepezil 10mg QD | Panel B: MK-1167 6mg QD + Donepezil 10mg QD | Panel B: Placebo to MK-1167 + Donepezil 10mg QD
Started | 12 | 4 | 9 | 3
Treated | 12 | 4 | 9 | 3
Panel A Participants Who Received 6mg of MK-1167 | 12 | 0 | 0 | 0
Panel A Participants Who Received 3mg of MK-1167 | 12 | 0 | 0 | 0
Completed | 10 | 4 | 8 | 3
Not Completed | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Serious Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-1167 + Donepezil 10mg QD | Panel A: Placebo to MK-1167 + Donepezil 10mg QD | Panel B: MK-1167 6mg QD + Donepezil 10mg QD | Panel B: Placebo to MK-1167 + Donepezil 10mg QD | Total
Number analyzed (Participants) | 12 | 4 | 9 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (8.2) | 63.5 (8.7) | 69.9 (8.6) | 75.3 (2.9) | 68.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 1 | 13
  Male | 6 | 1 | 6 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 4 | 2 | 12
  Not Hispanic or Latino | 8 | 2 | 5 | 1 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 3 | 0 | 11
  White | 6 | 2 | 6 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Panel A: Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC0-24) After Administration of 6mg of MK-1167
Description: AUC0-24 was defined as the area under the concentration-time curve of MK-1167 from time zero to 24 hours. Blood samples were collected at pre-specified intervals for the determination of AUC0-24. Per protocol, AUC0-24 was based on noncompartmental analysis, and a geometric mean AUC0-24 value was presented for Panel A participants after administration of 6mg of MK-1167.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel A randomized participants who received at least one dose of study treatment (6mg of MK-1167) and had at least one postdose data available for assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: μM*hour
Groups:
- Panel A: MK-1167 6mg QD + Donepezil 10mg QD: Participants received 6mg MK-1167 oral loading doses QD Days 1 to 7. Participants also receive 10mg oral Donepezil on Days -3 to 21.
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
μM*hour | 2.17 [1.22 to 3.84]

2. Secondary Outcome: Panel A: AUC0-24 After Administration of 3mg of MK-1167
Description: AUC0-24 was defined as the area under the concentration-time curve of MK-1167 from time zero to 24 hours. Blood samples were collected at pre-specified intervals for the determination of AUC0-24. Per protocol, AUC0-24 was based on noncompartmental analysis, and a geometric mean AUC 0-24 value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Days 8, 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel A randomized participants who received at least one dose of study treatment (3mg of MK-1167) and had at least one postdose data available for assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: μM*hour
Groups:
- Panel A: MK-1167 3mg QD + Donepezil 10mg QD: After an oral loading dose of 6mg MK-1167, participants received oral maintenance dose of 3mg MK-1167 QD Days 8 to 21. Participants also received 10mg oral Donepezil on Days -3 to 21.
Arm/Group | Panel A: MK-1167 3mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 12
μM*hour
  Day 8 | 8.70 [4.95 to 15.3]
  Day 21: number analyzed (Participants) | 10
  Day 21 | 8.08 [4.56 to 14.3]

3. Secondary Outcome: Panel B: AUC0-24 After Administration of 6mg of MK-1167
Description: AUC0-24 was defined as the area under the concentration-time curve of MK-1167 from time zero to 24 hours. Blood samples were collected at pre-specified intervals for the determination of AUC0-24. Per protocol, AUC0-24 was based on noncompartmental analysis, and a geometric mean AUC0-24 value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Days 1, 23, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment (6mg of MK-1167) and had at least one postdose data available for assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: μM*hour
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 9
μM*hour
  Day 1 | 2.48 [2.04 to 3.01]
  Day 23: number analyzed (Participants) | 8
  Day 23 | 22.2 [18.1 to 27.1]
  Day 31: number analyzed (Participants) | 8
  Day 31 | 22.9 [18.8 to 28.0]

4. Secondary Outcome: Panel A: Maximum Plasma Concentration (Cmax) After Administration of 6mg of MK-1167
Description: Cmax was defined as the maximum serum concentration of MK-1167 reached. Blood samples were collected at pre-specified timepoints for the determination of Cmax. Per protocol, Cmax was based on noncompartmental analysis, and a geometric mean Cmax value was presented for Panel A participants after administration of 6mg of MK-1167.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
μmol/Liter | 0.129 [0.0731 to 0.228]

5. Secondary Outcome: Panel A: Cmax After Administration of 3mg of MK-1167
Description: Cmax was defined as the maximum serum concentration of MK-1167 reached. Blood samples were collected at pre-specified timepoints for the determination of Cmax. Per protocol, Cmax was based on noncompartmental analysis, and a geometric mean Cmax value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Days 8, 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Panel A: MK-1167 3mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 12
μmol/Liter
  Day 8 | 0.434 [0.247 to 0.761]
  Day 21: number analyzed (Participants) | 10
  Day 21 | 0.413 [0.234 to 0.729]

6. Secondary Outcome: Panel B: Cmax After Administration of 6mg of MK-1167
Description: Cmax was defined as the maximum serum concentration of MK-1167 reached. Blood samples were collected at pre-specified timepoints for the determination of Cmax. Per protocol, Cmax was based on noncompartmental analysis, and a geometric mean Cmax value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Days 1, 23, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 9
μmol/Liter
  Day 1 | 0.145 [0.121 to 0.174]
  Day 23: number analyzed (Participants) | 8
  Day 23 | 1.11 [0.919 to 1.35]
  Day 31: number analyzed (Participants) | 8
  Day 31 | 1.14 [0.941 to 1.38]

7. Secondary Outcome: Panel A: Plasma Concentration at 24 Hours (C24) After Administration of 6mg of MK-1167
Description: C24 was defined as the serum concentration of MK-1167 reached at 24 hours. Blood samples were collected at pre-specified timepoints for the determination of C24. Per protocol, C24 was based on noncompartmental analysis, and a geometric mean C24 value was presented for Panel A participants after administration of 6mg of MK-1167.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
μmol/Liter | 0.0902 [0.0500 to 0.163]

8. Secondary Outcome: Panel A: C24 After Administration of 3mg of MK-1167
Description: C24 was defined as the serum concentration of MK-1167 reached at 24 hours. Blood samples were collected at pre-specified timepoints for the determination of C24. Per protocol, C24 was based on noncompartmental analysis, and a geometric mean C24 value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Days 8, 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel A randomized participants who received at least one dose of study treatment (3mg MK-1167) and had at least one postdose data available for assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Panel A: MK-1167 3mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 12
μmol/Liter
  Day 8 | 0.362 [0.203 to 0.647]
  Day 21: number analyzed (Participants) | 10
  Day 21 | 0.313 [0.174 to 0.565]

9. Secondary Outcome: Panel B: C24 After Administration of 6mg of MK-1167
Description: C24 was defined as the serum concentration of MK-1167 reached at 24 hours. Blood samples were collected at pre-specified timepoints for the determination of C24. Per protocol, C24 was based on noncompartmental analysis, and a geometric mean C24 value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Days 1, 23, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 9
μmol/Liter
  Day 1 | 0.0917 [0.0731 to 0.115]
  Day 23: number analyzed (Participants) | 8
  Day 23 | 0.729 [0.576 to 0.922]
  Day 31: number analyzed (Participants) | 8
  Day 31 | 0.875 [0.691 to 1.11]

10. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 7 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Panel B: MK-1167 6mg QD+ Donepezil 10mg QD: Participants received 6mg MK-1167 oral doses QD Days 1 to 31. Participants also receive 10mg oral Donepezil on Days -3 to 31.
- Panel B: Placebo to MK-1167 + Donepezil 10mg QD: Participants received dose matched placebo to MK-1167 oral QD from Days 1 to 31. Participants also received 10mg oral Donepezil QD on Days -3 to 31.
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD | Panel A: MK-1167 3mg QD + Donepezil 10mg QD | Panel A: Placebo to MK-1167 + Donepezil 10mg QD | Panel B: MK-1167 6mg QD+ Donepezil 10mg QD | Panel B: Placebo to MK-1167 + Donepezil 10mg QD
Number analyzed (Participants) | 12 | 12 | 4 | 9 | 3
Participants | 3 | 5 | 2 | 6 | 0

11. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 4 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Panel A: MK-1167 6mg QD + Donepezil 10mg QD: Participants received 6 mg MK-1167 oral loading doses QD Days 1 to 7. Participants also received 10mg oral Donepezil on Days -3 to 21.
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD | Panel A: MK-1167 3mg QD + Donepezil 10mg QD | Panel A: Placebo to MK-1167 + Donepezil 10mg QD | Panel B: MK-1167 6mg QD + Donepezil 10mg QD | Panel B: Placebo to MK-1167 + Donepezil 10mg QD
Number analyzed (Participants) | 12 | 12 | 4 | 9 | 3
Participants | 0 | 0 | 0 | 1 | 0

12. Secondary Outcome: Panel A: Time to Maximum Plasma Concentration (Tmax) After Administration of 6mg of MK-1167
Description: Tmax was defined as time to the maximum concentration of MK-1167 reached. Blood samples were collected at pre-specified intervals for the determination of Tmax. Per protocol, Tmax was based on noncompartmental analysis, and a median Tmax value was presented for Panel A participants after administration of 6mg of MK-1167.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
hours | 1.54 [0.50 to 8.00]

13. Secondary Outcome: Panel A: Tmax After Administration of 3mg of MK-1167
Description: Tmax was defined as time to the maximum concentration of MK-1167 reached. Blood samples were collected at pre-specified intervals for the determination of Tmax. Per protocol, Tmax was based on noncompartmental analysis, and a median Tmax value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Days 8, 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: MK-1167 3mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 12
hours
  Day 8 | 6.00 [0.00 to 23.97]
  Day 21: number analyzed (Participants) | 10
  Day 21 | 4.01 [1.22 to 11.92]

14. Secondary Outcome: Panel B: Tmax After Administration of 6mg of MK-1167
Description: Tmax was defined as time to the maximum concentration of MK-1167 reached. Blood samples were collected at pre-specified intervals for the determination of Tmax. Per protocol, Tmax was based on noncompartmental analysis, and a median Tmax value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Days 1, 23, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 9
hours
  Day 1 | 1.08 [0.48 to 5.78]
  Day 23: number analyzed (Participants) | 8
  Day 23 | 4.03 [0.58 to 11.92]
  Day 31: number analyzed (Participants) | 8
  Day 31 | 2.97 [0.42 to 11.90]

15. Secondary Outcome: Panel A: Apparent Clearance (CL/F) After Administration of 3mg of MK-1167
Description: CL/F is the rate at which the MK-1167 is completely removed from plasma. Blood samples were collected at pre-specified intervals for the determination of CL/F. Per protocol, CL/F was based on noncompartmental analysis, and a geometric mean CL/F value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Day 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360 and 480 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Panel A: MK-1167 3mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
Liter/hour | 0.879 (166.9)

16. Secondary Outcome: Panel B: CL/F After Administration of 6mg of MK-1167
Description: CL/F is the rate at which the MK-1167 is completely removed from plasma. Blood samples were collected at pre-specified intervals for the determination of CL/F. Per protocol, CL/F was based on noncompartmental analysis, and a geometric mean CL/F value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Day 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360 and 480 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Liter/hour | 0.606 (32.3)

17. Secondary Outcome: Panel A: Apparent Terminal Half-Life (t1/2) After Administration of 3mg of MK-1167
Description: t1/2 is defined as the time required to divide plasma concentration of MK-1167 by half after reaching pseudo-equilibrium. Blood samples were collected at pre-specified intervals for the determination of t1/2. Per protocol, t1/2 was based on noncompartmental analysis, and a geometric mean t1/2 value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Day 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360 and 480 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Panel A: MK-1167 3 mg QD + Donepezil 10mg QD: After an oral loading dose of 6mg MK-1167, participants received oral maintenance dose of 3mg MK-1167 QD Days 8 to 21. Participants also received 10mg oral Donepezil on Days -3 to 21.
Arm/Group | Panel A: MK-1167 3 mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
hours | 194 (48.2)

18. Secondary Outcome: Panel B: t1/2 After Administration of 6mg of MK-1167
Description: t1/2 was defined as the time required to divide plasma concentration of MK-1167 by half after reaching pseudo-equilibrium. Blood samples were collected at pre-specified timepoints for the determination of t1/2. Per protocol, t1/2 was based on noncompartmental analysis, and a geometric mean t1/2 value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Day 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360 and 480 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
hour | 193 (40.4)

19. Secondary Outcome: Panel A: Apparent Volume of Distribution (Vz/F) After Administration of 3mg of MK-1167
Description: Vz/F was the apparent volume of distribution of MK-1167. Blood samples were collected at pre-specified intervals for the determination of Vz/F. Per protocol, Vz/F was based on noncompartmental analysis, and a geometric mean Vz/F value was presented for Panel A participants after administration of 3mg of MK-1167.
Time Frame: Day 21: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360 and 480 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Panel A: MK-1167 3mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 10
Liter | 246 (166.6)

20. Secondary Outcome: Panel B: Vz/F After Administration of 6mg of MK-1167
Description: Vz/F was the apparent volume of distribution of MK-1167. Blood samples were collected at pre-specified intervals for the determination of Vz/F. Per protocol, Vz/F was based on noncompartmental analysis, and a geometric mean Vz/F value was presented for Panel B participants after administration of 6mg of MK-1167.
Time Frame: Day 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360 and 480 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Liter | 169 (19.7)

21. Secondary Outcome: Panel B: Day 23 to Day 1 Accumulation Ratio of AUC0-24 After Administration of 6mg of MK-1167
Description: Blood samples were collected at pre-specified timepoints to determine AUC0-24 on Days 1 and 23. AUC0-24 was defined as the area under the concentration-time curve of MK-1167 from time zero to 24 hours. Accumulation ratio of MK-1167 Day 23 to Day 1 was calculated as Day 23 AUC0-24/Day 1 AUC0-24.
Time Frame: Days 1, 23: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment and had AUC0-24 data available for assessment on Day 1 and Day 23.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Ratio | 8.95 [7.80 to 10.27]

22. Secondary Outcome: Panel B: Day 31 to Day 1 Accumulation Ratio of AUC0-24 After Administration of 6mg of MK-1167
Description: Blood samples were collected at pre-specified timepoints to determine AUC0-24 on Days 1 and 31. AUC0-24 was defined as the area under the concentration-time curve of MK-1167 from time zero to 24 hours. Accumulation ratio of MK-1167 Day 31 to Day 1 was calculated as Day 31 AUC0-24/Day 1 AUC0-24.
Time Frame: Days 1, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment and had AUC0-24 data available for assessment on Day 1 and Day 31.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Ratio | 9.26 [8.08 to 10.62]

23. Secondary Outcome: Panel B: Day 23 to Day 1 Accumulation Ratio of Cmax After Administration of 6mg of MK-1167
Description: Blood samples were collected at pre-specified timepoints to determine Cmax on Days 1 and 23. Cmax was defined as the maximum serum concentration of MK-1167 reached. Accumulation ratio of MK-1167 Day 23 to Day 1 was calculated as Day 23 Cmax/Day 1 Cmax.
Time Frame: Days 1, 23: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment and had at Cmax data available for assessment on Day 1 and Day 23.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Ratio | 7.69 [6.46 to 9.16]

24. Secondary Outcome: Panel B: Day 31 to Day 1 Accumulation Ratio of Cmax After Administration of 6mg of MK-1167
Description: Blood samples were collected at pre-specified timepoints to determine Cmax on Days 1 and 31. Cmax was defined as the maximum serum concentration of MK-1167 reached. Accumulation ratio of MK-1167 Day 31 to Day 1 was calculated as Day 31 Cmax/Day 1 Cmax.
Time Frame: Days 1, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment and had at Cmax data available for assessment on Day 1 and Day 31.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Ratio | 7.88 [6.62 to 9.38]

25. Secondary Outcome: Panel B: Day 23 to Day 1 Accumulation Ratio of C24 After Administration of 6mg of MK-1167
Description: Blood samples were collected at pre-specified timepoints to determine C24 on Days 1 and 23. C24 was defined as the serum concentration of MK-1167 reached at 24 hours. Blood samples were collected at pre-specified timepoints for the determination of C24. Accumulation ratio of MK-1167 Day 23 to Day 1 was calculated as Day 23 C24/Day 1 C24.
Time Frame: Days 1, 23: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment and had C24 data available for assessment on Day 1 and Day 23.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Ratio | 7.94 [6.64 to 9.50]

26. Secondary Outcome: Panel B: Day 31 to Day 1 Accumulation Ratio of C24 After Administration of 6mg of MK-1167
Description: Blood samples were collected at pre-specified timepoints to determine C24 on Days 1 and 31. C24 was defined as the serum concentration of MK-1167 reached at 24 hours. Blood samples were collected at pre-specified timepoints for the determination of C24. Accumulation ratio of MK-1167 Day 31 to Day 1 was calculated as Day 31 C24/Day 1 C24.
Time Frame: Days 1, 31: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: All Panel B randomized participants who received at least one dose of study treatment and had C24 data available for assessment on Day 1 and Day 31.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Panel B: MK-1167 6mg QD + Donepezil 10mg QD
Number analyzed (Participants) | 8
Ratio | 9.54 [7.97 to 11.40]

ADVERSE EVENTS:
Time Frame: Up to approximately 25 weeks
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) include all randomized participants who received ≥1 dose of study drug. Per protocol, Panel A: Placebo to MK-1167 + Donepezil 10mg QD arm was reported combined as dose matched placebo.
Groups:
- Panel A: MK-1167 6mg QD + Donepezil 10mg QD: Participants received 6mg MK-1167 oral loading doses QD Days 1to 7. Participants also received 10mg oral Donepezil on Days -3 to 21.
Arm/Group | Panel A: MK-1167 6mg QD + Donepezil 10mg QD | Panel A: MK-1167 3mg QD + Donepezil 10mg QD | Panel A: Placebo to MK-1167 + Donepezil 10mg QD | Panel B: MK-1167 6mg QD + Donepezil 10mg QD | Panel B: Placebo to MK-1167 + Donepezil 10mg QD
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/4 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/4 | 1/9 | 0/3
Other Adverse Events (participants affected / at risk) | 3/12 | 5/12 | 2/4 | 6/9 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-1167 6mg QD + Donepezil 10mg QD (N=12) | Panel A: MK-1167 3mg QD + Donepezil 10mg QD (N=12) | Panel A: Placebo to MK-1167 + Donepezil 10mg QD (N=4) | Panel B: MK-1167 6mg QD + Donepezil 10mg QD (N=9) | Panel B: Placebo to MK-1167 + Donepezil 10mg QD (N=3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-1167 6mg QD + Donepezil 10mg QD (N=12) | Panel A: MK-1167 3mg QD + Donepezil 10mg QD (N=12) | Panel A: Placebo to MK-1167 + Donepezil 10mg QD (N=4) | Panel B: MK-1167 6mg QD + Donepezil 10mg QD (N=9) | Panel B: Placebo to MK-1167 + Donepezil 10mg QD (N=3)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Any information identified by the Sponsor as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT06285240/Prot_SAP_000.pdf